CLINICAL TRIAL: NCT02795221
Title: Observative and Community Study, Using Nailfold Video-capillaroscopy in Order to Assess the Prevalence of Pathological Changes in the Capillaries in First Grade Family Members of Patient Diagnosed With Systemic Sclerosis
Brief Title: NVC Test in Order to Assess Pathological Changes in Family Members of Patient Diagnosed With SSc
Acronym: SSc NVC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, Head of Internal Medicine, Meir Medical Center
Other Study IDs: SSC-CAPI2016
Record Dates: First submitted 2016-06-05; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: According to the IRB Approval

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Systemic sclerosis (SSc) is multisystem autoimmune disease of unknown etiology. It's characterized by activation of immune system, microvascular changes and intimal proliferation.

The EULAR/ACR 2013 criteria for the classification of SSc will help identify SSC patients before fibrosis of internal organs and will allow early treatment.

Patient with RP, SSc-related autoAb, anti-topoisomerase I (SCL-70), anti-centromere autoAb, anti-RNApolymerase III, abnormal nailfold capillaries and puffy hands would have SSc.

The OR of abnormal capillaroscopy for subsequent development of SSc can reach 163 with positive predictive value of 52% and negative predictive value of 99% .Some studies found that preclinical internal organ involvement in pre-scleroderma patients, DLCO<80% was detected in 11/32 patients with RP plus SSc-associated autoAb plus SSc-type nailfold capillary changes.

The heritability of SSc was considered controversial in the, largest published SSc .Twin study, which in general suggested a modest genetic contribution to the Phenotype .Nevertheless, this study included only 42 sets of twins, and it should Be considered that, in a family study of 703 cases, an affected first-degree relative Increased the risk of SSc 13 times compared to the general population . Moreover, having an affected sibling increased SSc risk by 15 times , and there Was a remarkable concordance of auto antibodies between SSc twins . Additionally, recent analyses have shown that the standardized incidence ratio of SSc seemed to be less than those observed in autoimmune diseases (ADs) such as Rheumatoid arthritis or Ankylosing Spondylitis, but similar to those observed for Hashimoto, thyroiditis or psoriasis. In addition, SSc prevalence, clinical Outcomes and autoantibody profiles have been reported to vary depending on Patient ancestry Therefore, the role of genetic factors in SSc susceptibility can now be considered solidly established.

A positive family history of SSc appears to confer a risk that is at least 10-16-fold Higher than normal for SSc in first-degree relatives and 10-27-fold higher than Normal for SSc in siblings, and thus represents the strongest susceptibility factor Yet reported for this disease .

DETAILED DESCRIPTION:
Participates- 400 participates, males and females, 3-80 years old Study Plan

1. Review of trial method
2. Signing informed consent
3. Video-capillaroscopy
4. Questioning
5. Conclusions
6. Only for pathological findings-blood exams and follow-up at rheumatology clinic
7. Analysis of entire data
8. Final report Timeliness- After E.C Approvals- 2 years. Confidentiality & Privacy - As common in clinical trials, according to GCP and MOH guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patient hereby declare that he\she agree to participate the clinical trial, as detailed in the Informed Consent and sign the Informed Consent.
2. Patient is first Grade family member to systemic sclerosis patient.

Exclusion Criteria:

1. Patient refuses to sign Informed Consent.
2. Patient isn't first Grade family member to systemic sclerosis patient.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: first Grade family member to systemic sclerosis patient.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The Prevalence of abnormal nailfold capillaroscopy on First Grade Family relatives of patients with Systemic sclerosis | 1 year

IPD SHARING:
Plan to Share IPD: No
Principal investigator initiates